CLINICAL TRIAL: NCT06234657
Title: Effectiveness of Telerehabilitation on the Performance of Post-stroke Patients' Daily Living Activities and Evaluation of Satisfaction in Post-stroke Patients in Vietnam
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Science Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Doan Nguyen, Lecturer, University of Science Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversitySHCMC
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Telerehabilitation; Acute Stroke
Keywords: Stroke; Telerehabilitation
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The telerehabilitation program for stroke patients is provided via a remote system with caregiver support during 3 months
Masking Description: Outcomes Assessor will be randomly assigned to online interview the patient and caregiver (this person does not know and have previously treated the patient)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation for stroke patient (Experimental)
  Interventions: Behavioral: Telerehabilitation for stroke patient

INTERVENTIONS:
Behavioral: Telerehabilitation for stroke patient — The subjects of the study were intervened by telerehabilitation through video instructions and online group training via Online meeting software. The content of the intervention program included upper limb exercises, transfer, and ambulation functions. This training program was designed based on the clinical practice guidelines for post-stroke physiotherapy management from the United States Department of Veterans Affairs and the guidelines for the diagnosis, and treatment of rehabilitation stroke patients of the Vietnam Ministry of Health. The training results of the subjects will be evaluated by the Barthel Index

SUMMARY:
This study aims to evaluate the efficacy of telerehabilitation on stroke patients' capability to perform ADLs after three months of telerehabilitation intervention. Additionally, the investigators also conducted a survey on the satisfaction of patients after telerehabilitation

DETAILED DESCRIPTION:
The performance of stroke patients' daily living activities (ADLs) is severely affected because of hemiplegia. The consequences of stroke on patients can lead to a financial and welfare burden on society. Thus, it is vital to provide a rehabilitation program to enhance patients' performance in ADLs and help them become more independent. This study aims to evaluate the efficacy of telerehabilitation on stroke patients' capability to perform ADLs after three months of telerehabilitation intervention. Additionally, the investigators also conduct a survey on the satisfaction of patients after telerehabilitation. The investigators will recruit 32 stroke patients from five hospitals in Vietnam. All subjects will be provided the three-month treatment that includes video-based rehabilitation and the online meeting section. The investigators will use the Barthel Index (BI) to evaluate the intervention and use the Paired T-test to review the results. Evaluation of the satisfaction of stroke patients with telerehabilitation is conducted by Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ).

ELIGIBILITY:
Inclusion Criteria:

* Age: Over 18 years old
* Diagnosis: First stroke
* Stroke Severity: National Institutes of Health Stroke Scale (NIHSS) score between 5 and 15 (moderate impairment)
* Support System: Has a caregiver available during the research process
* Technology Access: Possesses a smartphone or computer with internet connection and online meeting application capabilities

Exclusion Criteria:

- Existing Conditions: Severe cognitive impairment, sensory impairment, language disorder, or musculoskeletal diseases limiting motor function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
The ability to perform several activities of daily living will be assess by Barthel Index (BI) | The patient was assessed using the BI scale at three time points: at the start of the study (discharge), one month after intervention and three months after the intervention
  Barthel Index (BI) is a scale that measures the ability to perform several activities of daily living. It consists of 10 items with a total score of 0 (lowest ability) to 100 (highest ability) . The 10 items of the scale refer to the patient's ability to eat, perform personal hygiene, bathe, dress, get on and off the toilet, control the bladder, control the bowels, move from a wheelchair to a bed and back, walk, and climb stairs.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided
To ensure participant confidentiality, all information will be encrypted and anonymized. Research results will be used for scientific purposes only.